CLINICAL TRIAL: NCT01425970
Title: A Phase II, Randomized, Multi-center, Two Part Study of the Safety and Efficacy of Double-blind, Placebo-controlled INX-08189 in Adjunctive Treatment With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Study Part A, and Open-label INX-08189 in Adjunctive (Interferon Free) Treatment With Daclatasvir and/or Ribavirin (Copegus®) in Study Part B, in Chronically-infected HCV Genotype 2 and 3 Treatment-naive Subjects
Brief Title: Chronically-infected HCV Genotype 2 and 3 Treatment-naive Subjects: Part A: Safety and Efficacy of INX-08189 With Peg IFN Alfa-2a and Ribavirin. Part B: INX-08189 in Interferon Free Treatment With Daclatasvir and/or Ribavirin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of study was due to safety reasons
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI472-003; INH-189-003 (Other: INH-189-003)
Record Dates: First submitted 2011-08-25; First posted 2011-08-30 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C
Keywords: Inhibitex; Chronic Hepatitis; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic | interventions — BMS-986094; peginterferon alfa-2a; Ribavirin; daclatasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 25 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin (Experimental): PART A Arm 1
  Interventions: Drug: INX-08189; Biological: Pegylated interferon alfa-2a; Drug: Ribavirin
- 50 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin (Experimental): PART A Arm 2
  Interventions: Drug: INX-08189; Biological: Pegylated interferon alfa-2a; Drug: Ribavirin
- 100 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin (Experimental): PART A Arm 3
  Interventions: Drug: INX-08189; Biological: Pegylated interferon alfa-2a; Drug: Ribavirin
- Placebo + Pegylated interferon alfa-2a + Ribavirin (Placebo Comparator): PART A Arm 4
  Interventions: Drug: Placebo matching with INX-08189; Biological: Pegylated interferon alfa-2a; Drug: Ribavirin
- 100 mg INX-08189 + Ribavirin (Experimental): PART B Arm 1
  Interventions: Drug: INX-08189; Drug: Ribavirin
- 200 mg INX-08189 + Ribavirin (Experimental): PART B Arm 2
  Interventions: Drug: Ribavirin; Drug: INX-08189
- Daclatasvir + INX-08189 100 mg (Experimental): PART B Arm 3
  Interventions: Drug: INX-08189; Drug: Daclatasvir
- Daclatasvir + INX-08189 200 mg (Experimental): PART B Arm 4
  Interventions: Drug: INX-08189; Drug: Daclatasvir
- Daclatasvir + INX-08189 50 mg + Ribavirin (Experimental): PART B Arm 5
  Interventions: Drug: INX-08189; Drug: Ribavirin; Drug: Daclatasvir

INTERVENTIONS:
Drug: INX-08189 — Tablet, Oral, 25 mg, Once daily (QD), 12 weeks
  Arms: 25 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin
Drug: INX-08189 — Tablet, Oral, 50 mg, Once daily (QD), 12 weeks
  Arms: 50 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; Daclatasvir + INX-08189 50 mg + Ribavirin
Drug: INX-08189 — Tablet, Oral, 100 mg, Once daily (QD), 12 weeks
  Arms: 100 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; 100 mg INX-08189 + Ribavirin; Daclatasvir + INX-08189 100 mg
Drug: Placebo matching with INX-08189 — Tablet, Oral, 0 mg, Once daily (QD), 12 weeks
  Arms: Placebo + Pegylated interferon alfa-2a + Ribavirin
Biological: Pegylated interferon alfa-2a — Syringe, Subcutaneous injection, 180 μg, Once per week, 12 weeks
  Arms: 100 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; 25 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; 50 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; Placebo + Pegylated interferon alfa-2a + Ribavirin
Drug: Ribavirin — Tablet, Oral, 500 or 600 mg weight dependent, Twice daily (BID), 12 weeks
  Arms: 100 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; 100 mg INX-08189 + Ribavirin; 200 mg INX-08189 + Ribavirin; 25 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; 50 mg INX-08189 + Pegylated interferon alfa-2a + Ribavirin; Daclatasvir + INX-08189 50 mg + Ribavirin; Placebo + Pegylated interferon alfa-2a + Ribavirin
Drug: INX-08189 — Tablet, Oral, 200 mg, QD, 12 weeks
  Arms: 200 mg INX-08189 + Ribavirin; Daclatasvir + INX-08189 200 mg
Drug: Daclatasvir — Tablet, Oral, 60 mg, QD, 12 weeks
  Other Names: BMS-790052
  Arms: Daclatasvir + INX-08189 100 mg; Daclatasvir + INX-08189 200 mg; Daclatasvir + INX-08189 50 mg + Ribavirin

SUMMARY:
Part A: The purpose of this study is to evaluate the safety and tolerability of INX-08189 and placebo with Peginterferon alfa-2a and Ribavirin during 12 weeks of treatment

Part B: The purpose of this study is to evaluate the safety and tolerability of INX-08189 with Ribavirin or INX-08189 with Daclatasvir or INX-08189 with Daclatasvir and Ribavirin

DETAILED DESCRIPTION:
Data Monitoring Committee is appointed for Part A only

Masking: Part A of this study is Double blind and the Part B is Open Label

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

Amendment 4: Genotype 1, 10 subjects at site 401.

* Males and females, 18 to 65 years of age inclusive with a body mass index (BMI) of at least 18 kg/m2 but not exceeding 36 kg/m2
* Diagnosed with chronic HCV at least 6 months prior to Visit 1 with medical documentation (e.g., prior PCR result, prior liver biopsy, prior genotyping, etc.), with a positive HCV viral load of at least 50,000 IU/mL at Visit 1 (screening) as measured by quantitative PCR
* Chronic genotype 2 or 3 HCV infection (per polymerase chain reaction [PCR] methodology)
* HCV treatment-naïve where "treatment-naïve" is defined as no prior treatment with IFN alfa 2a or 2b, Pegylated IFN alfa-2a, Ribavirin, or any HCV direct-acting anti-viral drugs
* Liver biopsy consistent with chronic HCV infection but with a classification of non-cirrhotic (and without classification of 'transition to cirrhosis or borderline cirrhosis') as judged by a pathologist (defined as Knodell ≤ 3, Metavir ≤ 2, Ishak ≤ 4, or Batts &Ludwig ≤ 2 ) within the last two years and before Visit 2 (biopsy can be done after Visit 1 and before Visit 2, within the screening period)
* Negative urine drug screen for drugs of abuse and methadone (via central lab-provided dipstick at site) at screening (Visit 1) (note: subjects with a valid prescription for a drug which can be abused [e.g., benzodiazepine, opiates] can be enrolled on the judgment of the investigator)
* Females will have a negative serum beta human chorionic gonadotropin (βHCG) pregnancy test at screening and a negative urine dipstick pregnancy test on Study Day 0 (visit 2)
* Agreement by both female subjects of childbearing potential and male subjects (who have not been surgically sterilized) to practice an acceptable method of birth control, which includes at least one barrier during the study and for at least 6 months after the cessation of treatment. Surgical sterilization of either the female or the male partner must have occurred at least 6 months prior to the first dose and females must be post-menopausal for 2 years to be considered of non-child-bearing potential. Acceptable contraceptive methods include one of the following: Oral and implantable hormonal contraceptives by the female partner for at least 3 months prior to the first dose of Study Drug with additional use of a barrier method, IUD in place for at least 6 months prior to first dose with additional use of barrier method. Acceptable barrier methods include either diaphragm with spermicide, and condom with spermicide. (Note: Abstinence is not an acceptable method of birth control, subjects who indicate sexual inactivity must agree to utilize an acceptable method of birth control in the event of sexual activity)
* Willing and able to complete all study visits and procedures, and able to effectively communicate with the investigator and other testing center personnel
* Signed informed consent form (ICF) executed prior to protocol screening assessments

Exclusion Criteria:

* Signs or symptoms of decompensated liver disease such as variceal bleeding, ascites, hepatic encephalopathy, active jaundice defined by an indirect bilirubin > 2, Alanine transaminase (ALT) or Aspartate aminotransferase (AST) laboratory values ≥ 10 times the upper limit of normal, or other evidence of decompensated liver disease, or hepatocellular carcinoma
* Chronic liver disease other than HCV not limited to Hepatitis B virus (HBV) [positive test for hepatitis B surface antigen (HBsAg)], hemochromatosis, auto-immune hepatitis, alcoholic liver disease or non-alcoholic fatty liver disease
* History of liver transplantation
* Co-infection with Human immunodeficiency virus (HIV) [positive test for anti-HIV Ab] or use of didanosine
* History of a heart attack, cardiac ischemia, heart disease, clinically symptomatic cardiac abnormalities, or blood clots, based on medical history or apparent on physical exam
* QTcF interval at Visit 1 of greater than or equal to 450 ms by Fridericia's correction, or a personal or family history of Torsades de Pointe
* History or presence of sarcoidosis or pancreatitis
* History or presence of severe pulmonary function impairment including severe (> GOLD stage III) chronic obstructive pulmonary obstructive disease, and moderate to severe asthma
* Uncontrolled diabetes mellitus as evidenced by HbA1C ≥ 8.5% at screening (Visit 1)
* Use of the following medications concurrently or within the 30 days prior to Screening (Visit 1) associated with QT prolongation: macrolides, antiarrhythmic agents, azoles, fluoroquinolones, and tricyclic anti-depressants (specifically excluded medication will be listed in protocol Section 6.8)
* Use of immunosuppressive or immune-modulating agents (including azathioprine, corticosteroids and immunosuppressive agents) or presence of an immunologically-mediated autoimmune disease (other than asthma) or history of solid organ or bone marrow transplantation (note: inhaled steroids for mild/moderate asthma and topical steroid for minor skin conditions allowed and washout period for per Oral (PO)/Intramuscular (IM)/ Intravenous (IV) corticosteroid use is 8 weeks; washout periods for other immunosuppressives determined by Medical Monitor)
* Use of strong CYP3A4-inhibiting protease inhibitors (specifically Atazanavir, Indinavir, Nelfinavir, Saquinavir, and Ritonavir), strong CYP3A4 inhibitors (specifically Clarithromycin, Itraconazole, Ketoconazole, Nefazodone, Telithromycin), or strong CYP3A4 inducers (specifically Rifampin, Efavirenz, Etravirine, Phenobarbital, Phenytoin, and Carbamazepine)
* Absolute neutrophil count of < 1800 cells/mm3, or platelet count < 130,000 cells/mm3, or hemoglobin < 12 g/dl for women and < 13 g/dl for men, or a history of anemia, sickle cell anemia, or thalassemia; (note: if baseline value within 5% of minimum qualifying value, one re-test allowed for the purpose of qualifying for study)
* A history or presence of abnormal thyroid function that is not adequately controlled [defined as Thyroid-stimulating hormone (TSH) levels less than 0.8 x lower limit of normal (LLN) or greater than 1.2 x the upper limit of normal (ULN)]
* Creatinine clearance < 50 mL/minute, serum creatinine concentration ≥ 1.5 times the ULN, or albumin ≤ 3 g/dl
* Presence or history of bipolar disorder, schizophrenia, psychosis, or unstable psychiatric condition, or hospitalization for psychiatric condition, or suicide attempt. (Note: Subjects with psychiatric conditions need to be adequately treated and on stable doses of appropriate medications for at least 3 months prior to Visit 1. History of suicidal ideation within prior 3 months is exclusionary)
* Any malignancy within the last 5 years other than treated cervical carcinoma in situ or treated basal cell carcinoma with no more than 20% risk of recurrence within 2 years
* Alcohol abuse by the assessment of the investigator within the past 2 years or an alcohol use pattern that will interfere with the study conduct
* Drug abuse by the assessment of the investigator within the last six months
* Pregnancy, current lactation in female subjects, or male subjects with partners who are pregnant, or females intending to become pregnant
* Major surgery within 30 days prior to Visit 1
* Participation in another clinical trial of an investigational drug or device within 6 months prior to Visit 1 unless that prior participation involved exposure only to placebo by clear and available documentation
* Donation of blood or plasma within 30 days prior to Visit 1 (not including routine laboratory assessments)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Part A: Change in Hepatitis C Viral Load Measurements at protocol specific timepoints | Weeks -6, 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 28, 36, 48
Part B: proportion of subjects with SVR defined as HCV RNA ≤ LOQ (Limit of Quantitation) | At treatment weeks 12
  * SVR = Sustained virologic response
  * HCV RNA = Hepatitis C virus ribonucleic acid
Part B: proportion of subjects with SVR defined as HCV RNA ≤ LOQ | Post treatment week 12
Safety assessments is measured by Physical Exams, vital signs, laboratory assessments, ECGs, pregnancy test, viral resistance testing, adverse event assessment | up to 1 year

SECONDARY OUTCOMES:
Proportion of subjects with RVR (Rapid Virologic Response), undetectable HCV RNA | At treatment weeks 4
Proportion of subjects with Complete EVR (Early Virologic Response), undetectable HCV RNA | At treatment weeks 12
Proportion of subjects with Extended RVR | At treatment weeks 4 and 12
Proportion of subjects with SVR24 | Post treatment week 24
  SVR24 = sustained virologic response at 24 weeks after the cessation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (6):
  - Acri Phase One, Anaheim, California
  - Scripps Health Dba Scripps Clinical Research Services, La Jolla, California
  - Quest Clinical Research, San Francisco, California
  - Kansas City Cancer Centers, Llc., Kansas City, Missouri
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Alamo Medical Research, San Antonio, Texas

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx